CLINICAL TRIAL: NCT02289703
Title: An Open-label Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of a Single Dose of Rivaroxaban in Subjects With End-Stage Renal Disease (ESRD) on Maintenance Hemodialysis
Brief Title: A Pharmacokinetics, Pharmacodynamics and Safety Study of Single Dose of Rivaroxaban in Participants With End-Stage Renal Disease (ESRD) on Maintenance Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR105711; RIVAROXCRF1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: End-Stage Renal Disease
Keywords: End-Stage Renal Disease; Healthy; Rivaroxaban; BAY 59-7939; JNJ-39039039; Xarelto; Hemodialysis; Blood Coagulation; Pharmacokinetics
MeSH Terms: conditions — Kidney Failure, Chronic; Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Participants with end-stage renal disease (ESRD), will receive a single 15-milligram (mg) oral dose of rivaroxaban in Treatment Period 1 on Day 1, administered 2 hours before the start of a 4-hour hemodialysis session followed 7 to 14 days later by Treatment Period 2 wherein a single 15-mg oral dose of rivaroxaban will be given 3 hours after the completion of a 4-hour hemodialysis session on Day 1.
  Interventions: Drug: Rivaroxaban 15 mg
- Group B (Experimental): Healthy control participants matching to 'Group A' participants, will receive a single 15-mg oral dose of rivaroxaban on Day 1.
  Interventions: Drug: Rivaroxaban 15 mg

INTERVENTIONS:
Drug: Rivaroxaban 15 mg — Single oral dose of rivaroxaban 15-mg tablet on Day 1 of each of the treatment periods.
  Other Names: JNJ-39039039; BAY 59-7939; Xarelto

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (the study of the way a drug enters and leaves the blood and tissues over time) and pharmacodynamics (the way a drug may change body function) of a single 15-milligram (mg) dose of rivaroxaban in both healthy participants with a creatinine clearance (CLcr) greater than equal to (>=) 80 milliliter per minute (mL/min) and clinically stable participants with end-stage renal disease (ESRD) on maintenance hemodialysis (a method used to remove waste material from the blood when the kidneys are unable to do so).

DETAILED DESCRIPTION:
This is an open-label (participants and researchers are aware about the treatment, participants are receiving), single-dose, single-center, parallel group (a medical research study comparing the response in 2 or more groups of participants receiving different interventions) study. This study consists of a Screening Period (within 21 days prior to admission into the study center on Day -1), followed by 2 treatment periods for ESRD participants (Group A) (Treatment Period 1: rivaroxaban will be administered 2 hours before the start of a 4-hour hemodialysis session on Day 1; Treatment Period 2: rivaroxaban will be administered 3 hours after the completion of a 4-hour hemodialysis session on Day 1), or 1 treatment period for healthy participants (Group B) (single oral dose of rivaroxaban will be administered on Day 1). Each treatment period will have duration of 4 days. For ESRD participants, the 2 treatments periods will be separated by a washout period of at least 7 days and a maximum of 14 days. The total study duration for ESRD participants is approximately 43 days. The total study duration for healthy participants is approximately 25 days. Blood samples will be collected to assess pharmacokinetic and pharmacodynamic parameters. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

A. All Participants:

- Body mass index (BMI = weight in kilogram [kg] divided by the square of height in meter [m]) between 18 and 38 kg/m^2, extremes included, and body weight not less than 50 kg

B. Additional Inclusion Criteria for ESRD Participants (Group A):

* Participants with end-stage renal disease (ESRD) requiring maintenance hemodialysis 2 or 3 times a week for at least 3 months prior to Screening
* Participants with clinically stable medical condition, consistent with ESRD, as judged by the investigator on the basis of the Screening physical examination, medical history, vital signs, 12-lead electrocardiogram (ECG), and results of clinical laboratory tests performed within 3 weeks of the first administration of study drug (unless judged to be clinically unimportant by the investigator or sponsor)
* Participants with diastolic blood pressure less than (<) 110 millimeter of mercury (mmHg) and/or systolic blood pressure <180 mmHg (at Screening only) recorded after 5 minutes rest in sitting position

C. Additional Inclusion Criteria for Healthy Matched Control Participants (Group B):

* Healthy Participants on the basis of Screening physical examination, medical history, vital signs, 12-lead ECG, and results of clinical laboratory tests performed within 3 weeks prior to the administration of study drug
* Participants with diastolic blood pressure <95 mmHg and/or systolic blood pressure <150 mmHg recorded after 5 minutes rest in sitting position
* Participants with normal renal function characterized as having creatinine clearance (CLcr) >80 mL/min by Cockcroft-Gault estimate

Exclusion Criteria:

* Participants with history of clinically significant medical illness prior to Screening including (but not limited to) chronic atrial fibrillation, hemodynamically significant valvular heart disease, heart failure (New York Heart Association Class >=II) within 6 months prior to the Screening visit, cardiac revascularization within 6 months including percutaneous transluminal coronary angioplasty or coronary artery bypass graft surgery, ischemic stroke within 6 months, previous intracranial hemorrhage at any time, anemia with a hemoglobin concentration <9 gram per deciliter (g/dL), or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participants diagnosed with current malignancy/active disease; (however, participants with clinically stable prostate cancer, basal cell carcinoma of the skin or who have not required antineoplastic treatment of previous cancers for at least one year are eligible)
* Participants with psychiatric disorders that would impair the participant's ability to participate or complete this study in the opinion of the investigator or the sponsor
* Participants with history of gastrointestinal disease (for example, Crohn's disease) which could result in impaired absorption of the study drugs
* Participants with any other disease or condition which could influence the physiological metabolic turnover of study drug (for example, endocrine diseases, febrile conditions, severe infections)
* Participants with history of significant hemorrhage and gastrointestinal ulceration within 6 months prior to the screening visit
* Participants with known primary coagulation disorders (for example, von Willebrand's disease, hemophilias)
* Participants with history of recurrent dialysis membrane thrombosis
* Participants with sensitivity to heparin
* Participants with dialysis for acute renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Rivaroxaban | Pre-dose up to 72 hrs post-dose
  The Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration-time Curve From Time Zero to Last Quantifiable Time (AUClast) of Rivaroxaban | Pre-dose up to 72 hrs post-dose
  The AUClast is the area under the plasma concentration-time curve from time zero to time of last quantifiable concentration.
Area Under the Plasma Concentration-time Curve From Time Zero to Extrapolated Infinite Time (AUCinfinity) of Rivaroxaban | Pre-dose up to 72 hrs post-dose
  The AUCinfinity is the area under the plasma concentration-time curve from time zero to extrapolated infinite time, calculated as the sum of AUClast and Clast/lambda(z), where AUClast is area under the plasma concentration-time curve from time zero to time of last quantifiable plasma concentration; Clast is the last observed quantifiable concentration; and lambda(z) is first-order rate constant associated with the terminal portion of the semilogarithmic drug concentration-time curve.

SECONDARY OUTCOMES:
Maximum Observed Effect (Emax) for Prothrombin Time (PT), Factor Xa (FXa) Inhibition and Anti-FXa | Pre-dose up to 72 hrs post-dose
  Maximum observed effect (Emax) for parameters: prothrombin time (PT), factor Xa (FXa) inhibition and anti-FXa, will be assessed.
Area Under the Dose-Response Curve for Prothrombin Time (PT), Factor Xa (FXa) Inhibition and Anti-FXa | Pre-dose up to 72 hrs post-dose
  The area under the dose-response curve for parameters: prothrombin time, FXa inhibition and anti-FXa, will be assessed.
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | Screening up to end of study (Group A: maximum up to 43 days, Group B: maximum up to 25 days) or up to early withdrawal
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Knoxville, Tennessee, United States

REFERENCES:
- See also: An Open-label Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of a Single Dose of Rivaroxaban in Subjects with End-Stage Renal Disease (ESRD) on Maintenance Hemodialysis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=8598&filename=CR105711_CSR%20Synopsis.pdf